CLINICAL TRIAL: NCT06810024
Title: Stroke Homecare and Recurrence Prevention
Acronym: SHARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Xuejun Yin, Prof, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAMS&PUMC-IEC-2025-008; 2021-RC330-004 (Other Grant/Funding Number: Chinese Academy of Medical Sciences)
Record Dates: First submitted 2025-01-21; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: stroke; home-based care
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervetnion group (Home-Based care group) (Experimental): Participants in this arm will receive a comprehensive home-based health care program designed to prevent stroke recurrence and enhance recovery. The intervention includes monitoring and management of stroke recurrence risk factors (e.g., blood pressure, blood sugar, cholesterol), functional rehabilitation, psychological health support, nutritional and lifestyle interventions, complication prevention, and caregiver empowerment. These interventions will be delivered over a 12-month period, and participants will be followed up at 6 and 12 months.
  Interventions: Combination Product: Home-based therapy
- Control group (standard care group) (Active Comparator): Participants in this arm will receive standard post-stroke care according to local clinical guidelines. This care may include outpatient visits for monitoring and medication management, inpatient rehabilitation services (e.g., physical, occupational, speech therapy), follow-up appointments with healthcare providers, and community-based rehabilitation services. Participants will be followed up at 6 and 12 months to assess stroke recurrence and recovery outcomes.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Combination Product: Home-based therapy — The home-based intervention includes the following modules:
  1. Management of Stroke Recurrence Risk Factors: Home-based monitoring and management of blood pressure, blood sugar, cholesterol, and medication adherence.
  2. Functional Rehabilitation and Daily Living Skills: Home-based physical therapy, rehabilitation exercises, and recovery of daily living skills.
  3. Psychological Health and Emotional Management: Home-based counseling and mental health support to address anxiety, depression, and stress.
  4. Nutritional and Lifestyle Interventions: At-home guidance on healthy eating, lifestyle changes, and behavior modification to reduce stroke recurrence.
  5. Risk and Complication Prevention: Home monitoring to prevent infections and other complications during recovery.
  6. Caregiver Empowerment: Home-based caregiver training and support to improve caregiving skills and reduce caregiver stress.
  Arms: Intervetnion group (Home-Based care group)
Other: Standard Care (in control arm) — The standard care intervention involves:
  Outpatient Visits: Routine follow-up visits to healthcare providers for stroke recovery monitoring, medication management, and adjustments.
  Inpatient Rehabilitation: Physical, occupational, and speech therapy delivered in hospital or rehabilitation centers, if required.
  Follow-up Appointments: Regular visits with stroke specialists and rehabilitation professionals for ongoing care.
  Arms: Control group (standard care group)

SUMMARY:
Background and Significance:

Stroke is the leading cause of death in China, placing a heavy burden on patients, families, and society. Despite advancements in acute stroke treatment, the recurrence rate remains high, and secondary prevention faces significant challenges. Current standard care does not fully address the diverse needs of stroke patients. Home-based health care (HBHC) offers a promising new intervention, providing continuous medical support, personalized lifestyle changes, and improved medication adherence, potentially reducing the risk of stroke recurrence.

Study Objectives and Hypotheses:

The study seeks to assess the impact of HBHC on reducing stroke recurrence, improving quality of life, enhancing physical function, addressing psychological health issues, and increasing medication adherence. Additionally, the study will explore the cost-effectiveness of HBHC in reducing medical resource utilization and preventing cardiovascular events. It is hypothesized that HBHC will effectively reduce stroke recurrence and improve overall health outcomes.

Study Design This study is a multicenter, randomized controlled trial designed to assess the effectiveness and cost-effectiveness of a home-based health care (HBHC) model in preventing recurrent strokes. A total of 1,614 stroke patients will be recruited from multiple regions in China and randomly assigned in a 1:1 ratio to either the intervention group or the control group. The intervention group will receive a comprehensive 12-month HBHC program that includes managing stroke recurrence risk factors, functional rehabilitation, daily living skills recovery, psychological health interventions, nutritional and lifestyle counseling, risk prevention, and caregiver empowerment. In contrast, the control group will receive standard post-stroke care and follow-up according to local guidelines. Both groups will undergo follow-up assessments at 6 and 12 months to evaluate stroke recurrence, quality of life, physical function, and psychological health. The study will span 2 years, with the primary outcome being the stroke recurrence rate within 12 months. Secondary outcomes include improvements in quality of life, physical function recovery, psychological health, medication adherence, cardiovascular events, and medical resource utilization. A process evaluation will also be conducted to assess the feasibility, adaptability, and implementation challenges of the HBHC model across different regions and patient populations.

Value and impact:

The findings will offer valuable insights into the feasibility and adaptability of HBHC across different regions and patient populations, contributing to the development of evidence-based strategies for improving long-term stroke management. Ultimately, this research will inform policy decisions, enhance clinical practice, and support the broader adoption of HBHC interventions to mitigate the burden of stroke and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosed with ischemic or hemorrhagic stroke within the past month
* Clinically stable, having completed acute phase treatment, and about to be discharged in a normal condition
* Physically able to receive home-based health care services
* Residing in a community where home-based health care is available
* Able to provide informed consent or have a legally authorized representative provide consent

Exclusion Criteria:

* Receiving more than one month of post-discharge care at a stroke rehabilitation center or community rehabilitation center
* Severe comorbidities (e.g., cancer, respiratory failure, severe infections) with a life expectancy of less than 6 months
* Severe cognitive impairment or mental illness affecting adherence to the intervention
* Currently participating in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1614 (Estimated)
Dates: Start 2025-02-27 (Estimated); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Stroke Recurrence Rate within 12 Months of Intervention | 12 months after the start of the intervention
  This outcome measures the occurrence of stroke recurrence in participants during the 12-month period following the start of the intervention. It aims to assess the effectiveness of the home-based health care intervention in reducing the risk of stroke recurrence compared to standard post-stroke care. Recurrence will be defined as a clinically confirmed stroke event (ischemic or hemorrhagic) occurring within 12 months of the intervention's initiation.

SECONDARY OUTCOMES:
Cardiovascular Events | 12 months after the start of the intervention
  This outcome measures the occurrence of cardiovascular events, including heart attacks, arrhythmias, and other major cardiovascular incidents, as confirmed by clinical doctors through electronic medical records, electrocardiograms, and imaging studies during the follow-up period.
All-Cause Mortality | 12 months after the start of the intervention
  This outcome tracks the occurrence of all-cause death during the study period, obtained through hospital records and death certificates.
Motor Function | 6 months and 12 months after the start of the intervention
  This outcome assesses changes in motor function using standardized scale such as the Modified Rankin Scale (mRS)
Motor Function assessed by Barthel Index | 6 months and 12 months after the start of the intervention
  This outcome assesses changes in motor function using standardized scale as the Barthel Index.
Cognitive Function | 6 months and 12 months after the start of the intervention.
  This outcome evaluates changes in cognitive function using assessments such as the Mini-Mental State Examination (MMSE).
Depression | 6 months and 12 months after the start of the intervention
  This outcome evaluates changes in depression levels using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a standardized tool for assessing the severity of depressive symptoms. The PHQ-9 score ranges from 0 to 27, with higher scores indicating worse depression severity.
Anxiety | 6 months and 12 months after the start of the intervention.
  This outcome assesses changes in anxiety levels using the Generalized Anxiety Disorder-7 (GAD-7) scale. The GAD-7 is a widely used tool for screening and measuring the severity of generalized anxiety disorder symptoms. The GAD-7 score ranges from 0 to 21, with higher scores indicating worse anxiety severity.
Quality of Life using the EQ-5D scale | 6 months and 12 months after the start of the intervention
  This outcome measures quality of life using the EQ-5D scale, which assesses various health dimensions such as mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Healthcare Utilization (Hospitalizations and Emergency Visits) | 12 months after the start of the intervention
  This outcome evaluates the frequency of hospitalizations and emergency visits during the study period, as documented in hospital electronic medical records, emergency department records, and patient-reported data, confirmed through follow-up visits.
Knowledge, Beliefs, and Behaviors Related to Stroke Recurrence Prevention | 12 months after the start of the intervention
  This outcome measures participants' knowledge, beliefs, and behaviors regarding stroke recurrence prevention, assessed through a structured survey questionnaire.

IPD SHARING:
Plan to Share IPD: Undecided
In this study, individual participant data (IPD) might not be shared due to concerns related to privacy and confidentiality. Since the study involves sensitive health information, including stroke diagnoses, rehabilitation progress, and psychological assessments, sharing IPD could potentially violate participant privacy or breach confidentiality agreements.